CLINICAL TRIAL: NCT07276087
Title: Physical and Psychosocial Parameters in Takayasu Arteritis and Behçet's Disease: A Comparative Study With Healthy Controls
Status: Recruiting | Type: Observational
Sponsor: ÖZLEM NUR TOK YAMAN (Other)
Collaborators: Pamukkale University (Other); Uşak University (Other); Alanya Alaaddin Keykubat University (Other)
Responsible Party: Sponsor-Investigator, ÖZLEM NUR TOK YAMAN, Lecturer , Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Alanya Alaaddin Keykubat University
Organization: Alanya Alaaddin Keykubat University (Other)
Other Study IDs: PAU-KAEK-2025-17
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Takayasu Arteritis; Behçet's Disease; Healthy Controls
Keywords: Takayasu arteritis; Behçet's disease; Systemic vasculitis; Muscle strength
MeSH Terms: conditions — Takayasu Arteritis; Behcet Syndrome; Systemic Vasculitis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Takayasu Arteritis Group: Participants diagnosed with Takayasu arteritis according to established clinical and imaging criteria.
  Interventions: Other: No intervention (observational study)
- Behçet's Disease Group: Participants diagnosed with Behçet's disease according to the International Study Group criteria.
  Interventions: Other: No intervention (observational study)
- Healthy Control Group: Age- and sex-matched healthy volunteers with no systemic or chronic disease.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — Participants will not receive any treatment or intervention. The study involves only physical and psychosocial assessments and questionnaires.

SUMMARY:
Systemic vasculitis refers to a group of rare diseases characterized by inflammation of blood vessel walls, which may cause ischemia and structural damage in various organs. Among large-vessel vasculitides, Takayasu arteritis primarily affects the aorta and its main branches, whereas Behçet's disease is a variable vessel vasculitis involving arteries and veins of all sizes. Both conditions can lead to multisystemic involvement and significantly impact physical and psychosocial health.

This observational, case-control study aims to compare multiple physical and psychosocial parameters among individuals with Takayasu arteritis, Behçet's disease, and healthy controls. Assessments will include respiratory and peripheral muscle strength, functional status, exercise capacity, body composition, quality of life, illness perception, and psychological well-being. Measurements will be conducted using standardized clinical tests (such as maximal inspiratory and expiratory pressures, handgrip and limb strength dynamometry, squat test, and six-minute walk test) and validated questionnaires (Health Assessment Questionnaire (HAQ), the Short Form-36 Health Survey (SF-36), the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L), and the Visual Analogue Scale (VAS)).

The study seeks to identify differences between groups and provide a comprehensive understanding of how systemic inflammation in Takayasu arteritis and Behçet's disease affects physical performance, quality of life, and psychosocial health. These findings may help guide physiotherapy, rehabilitation, and multidisciplinary management strategies for patients with systemic vasculitis.

DETAILED DESCRIPTION:
Systemic vasculitis represents a heterogeneous group of rare inflammatory diseases that affect blood vessel walls, potentially leading to ischemia, tissue damage, and multi-organ dysfunction. Among them, Takayasu arteritis (TAK) and Behçet's disease (BD) are chronic, relapsing vasculitides characterized by systemic inflammation and variable vessel involvement. These diseases may cause not only organ-specific pathology but also generalized effects on muscle strength, physical function, and psychosocial well-being.

Previous studies have reported reduced physical performance, fatigue, and impaired quality of life in patients with systemic vasculitis. However, there is limited evidence directly comparing physical and psychosocial parameters between individuals with Takayasu arteritis, Behçet's disease, and healthy controls. The current literature lacks a comprehensive approach addressing the multidimensional impact of these diseases on functional and psychological outcomes.

This observational, cross-sectional study aims to fill this gap by evaluating and comparing respiratory and peripheral muscle strength, functional capacity, quality of life, illness perception, and related psychosocial parameters among these three groups. Measurements will include maximal inspiratory and expiratory pressures, handgrip and limb muscle strength via digital dynamometry, functional tests such as the squat test and the six-minute walk test, and standardized self-reported questionnaires including the Health Assessment Questionnaire (HAQ), the Short Form-36 Health Survey (SF-36), the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L), and the Visual Analogue Scale (VAS).

The study is expected to provide a multidimensional understanding of how systemic inflammation in Takayasu arteritis and Behçet's disease affects physical and psychosocial functioning. The findings are anticipated to contribute to the literature by highlighting differences between disease groups and healthy controls and to guide future physiotherapy and rehabilitation strategies aimed at improving overall health and quality of life in individuals with systemic vasculitis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Takayasu Arteritis Group):

* Age 18 years or older.
* Diagnosis of Takayasu arteritis according to the American College of Rheumatology (ACR) classification criteria.
* Voluntary participation with written informed consent.

Inclusion Criteria (Behçet's Disease Group):

* Age 18 years or older.
* Diagnosis of Behçet's disease according to the International Study Group for Behçet's Disease criteria.
* Voluntary participation with written informed consent.

Inclusion Criteria (Healthy Control Group):

* Age 18 years or older.
* No history of systemic, rheumatologic, or chronic inflammatory disease.
* Voluntary participation with written informed consent.

Exclusion Criteria:

Exclusion Criteria (Patient Groups - Takayasu Arteritis and Behçet's Disease):

* Pregnancy.
* Presence of psychiatric disorder or ongoing psychiatric treatment.
* Cognitive impairment that may interfere with participation.
* Presence of neurological disease (e.g., hemiplegia, Parkinson's disease, multiple sclerosis, vertigo, epilepsy, etc.).
* History of any surgical operation within the past year.
* Coexisting rheumatic disease other than Takayasu arteritis or Behçet's disease.

Exclusion Criteria (Healthy Control Group):

* Pregnancy.
* Presence of psychiatric disorder or ongoing psychiatric treatment.
* Cognitive impairment that may interfere with participation.
* Presence of neurological disease (e.g., hemiplegia, Parkinson's disease, multiple sclerosis, vertigo, epilepsy, etc.).
* History of any surgical operation within the past year.
* History of rheumatologic or chronic inflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals aged 18 years and older who have been diagnosed with Takayasu arteritis or Behçet's disease and are being followed at the Rheumatology Department of Pamukkale University, as well as age- and sex-matched healthy volunteers without systemic, neurological, or musculoskeletal disease. All participants will provide written informed consent prior to inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral muscle strength | Single assessment (baseline only)
  Peripheral muscle strength will be assessed using the Commander Echo™ Muscle Testing Dynamometer (JTECH Medical, USA) for upper and lower extremities. Measurements will include quadriceps, biceps, and shoulder abductor muscle strength. The average of three trials will be recorded in kilograms.
Respiratory Muscle Strength | Single assessment (baseline only)
  Measured by maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using a portable electronic manometer (Micro Medical MicroMPM, UK).

SECONDARY OUTCOMES:
Functional Exercise Capacity-Six-Minute Walk Test (6MWT) | Single session at baseline
  Assessed by the Six-Minute Walk Test (6MWT), following standardized ATS/ERS guidelines. Distance walked will be recorded in meters.
Functional Status- Health Assessment Questionnaire | Single session at baseline
  Evaluated using the Health Assessment Questionnaire (HAQ). Scores range from 0 to 3, with higher scores indicating worse disability.
General Health Perception - Visual Analogue Scale (VAS) | Single assessment at baseline.
  General health perception will be assessed using the Visual Analogue Scale (VAS). The VAS consists of a 100 mm horizontal line anchored by "very good" at one end and "very poor" at the other. Participants are asked to mark a point on the line that best represents their perceived general health. The score is determined by measuring the distance in millimeters from the "very good" anchor to the participant's mark. Higher scores indicate worse perceived health status.
Quality of Life - Short Form-36 Health Survey (SF-36) | Single session at baseline
  The SF-36 (Short Form Health Survey) will assess health-related quality of life. Scores range from 0 to 100; higher scores indicate better health status.
Quality of Life - EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) | Single session at baseline.
  Quality of life will be assessed using the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L). The EQ-5D-5L includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each scored from 1 to 5, where higher scores indicate more severe problems. The instrument also includes a Visual Analogue Scale (VAS), on which participants rate their overall health from 0 (worst imaginable health) to 100 (best imaginable health). Higher VAS scores indicate better perceived health.
Illness Perception - Illness Perception Questionnaire (IPQ) | Single session at baseline
  Illness perception will be assessed using the Illness Perception Questionnaire (IPQ). Higher scores indicate stronger negative illness perceptions.
Fat Mass (kilograms) | Single session at baseline
  Measured via bioelectrical impedance analysis using the Polosmart PSC12 Prolife device. Recorded in kilograms.
Muscle Mass (kilograms) | Single session at baseline
  Measured via bioelectrical impedance analysis using the Polosmart PSC12 Prolife device. Recorded in kilograms.
Body Fat Percentage | Single session at baseline.
  Measured via bioelectrical impedance analysis using the Polosmart PSC12 Prolife device. Recorded as percentage of total body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided